CLINICAL TRIAL: NCT01149122
Title: Phase III Study of Gemcitabine/Oxaliplatin (GEMOX) With or Without Erlotinib in Unresectable, Metastatic Biliary Tract Carcinoma
Brief Title: Gemcitabine/Oxaliplatin (GEMOX) With or Without Erlotinib (Tarceva) in Advanced Biliary Tract Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-12-024
Record Dates: First submitted 2010-01-07; First posted 2010-06-23 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-01

CONDITIONS: Unresectable, Metastatic Biliary Tract Carcinoma
Keywords: unresectable, metastatic biliary tract carcinoma; Gemcitabine/Oxaliplatin (GEMOX); Erlotinib
MeSH Terms: interventions — gemcitabine-oxaliplatin regimen; Gemcitabine; Oxaliplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine/Oxaliplatin with Erlotinib (Active Comparator)
  Interventions: Drug: Gemcitabine/Oxaliplatin with Erlotinib (Tarceva)
- Gemcitabine/Oxaliplatin without Erlotinib (Active Comparator)
  Interventions: Drug: Gemcitabine/Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine/Oxaliplatin — GEMOX: (Gemcitabine 100 mg/㎡ over 100-min, Oxaliplatin 100 mg/㎡ over 2h) q (every) 2 weeks
  Arms: Gemcitabine/Oxaliplatin without Erlotinib
Drug: Gemcitabine/Oxaliplatin with Erlotinib (Tarceva) — GEMOX + Tarceva: (Gemcitabine 1000 mg/㎡ over 100-min, Oxaliplatin 100 mg/㎡ over 2h) q 2weeks; Tarceva 100 mg qd
  Arms: Gemcitabine/Oxaliplatin with Erlotinib

SUMMARY:
The purpose of this study is to determine whether Gemcitabine/Oxaliplatin (GEMOX) with or without Erlotinib (Tarceva) is effective in the treatment of unresectable, metastatic biliary tract carcinoma.

DETAILED DESCRIPTION:
This is a phase III study of Gemcitabine/Oxaliplatin (GEMOX) with or without Erlotinib in unresectable, metastatic biliary tract carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. histologically or cytologically confirmed adenocarcinoma of biliary tract
3. unresectable or metastatic
4. ECOG performance status of 0~2
5. measurable or evaluable lesion per RECIST criteria
6. adequate marrow, hepatic, renal and cardiac functions
7. no prior chemotherapy or molecularly targeted therapy for the advanced biliary carcinoma (prior adjuvant chemotherapy will be allowed if administered ≥ 6 months from the study entry)
8. provision of a signed written informed consent

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. active CNS metastases not controllable with radiotherapy or corticosteroids
4. known history of hypersensitivity to study drugs
5. prior exposure to EGFR tyrosine kinase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | every 6 weeks

SECONDARY OUTCOMES:
Safety profile | 24 months
Response rate | 24 months
Duration of response | 24 months
Time to progression | 24 months
Overall survival | 24 months
Correlative analyses: EGFR mutation, EGFR amplification, akt expression, EGFR polymorphism analyses | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ho yeong Lim, M.D,Ph.D, Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Jang KT, Lee SJ, Jang HL, Lee J, Park SH, Park YS, Lim HY, Kang WK, Park JO. Tumour shrinkage at 6 weeks predicts favorable clinical outcomes in a phase III study of gemcitabine and oxaliplatin with or without erlotinib for advanced biliary tract cancer. BMC Cancer. 2015 Jul 21;15:530. doi: 10.1186/s12885-015-1552-y. PMID 26189560
- [Derived] Lee J, Park SH, Chang HM, Kim JS, Choi HJ, Lee MA, Jang JS, Jeung HC, Kang JH, Lee HW, Shin DB, Kang HJ, Sun JM, Park JO, Park YS, Kang WK, Lim HY. Gemcitabine and oxaliplatin with or without erlotinib in advanced biliary-tract cancer: a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2012 Feb;13(2):181-8. doi: 10.1016/S1470-2045(11)70301-1. Epub 2011 Dec 20. PMID 22192731